CLINICAL TRIAL: NCT04576494
Title: Study of the Functional Effects of Nusinersen in 5q-spinal Muscular Amyotrophy Adults (SMA Type 2 or 3 Forms): a Multicenter Single-case Experimental Design in Multiple Baselines Across Subjects, Randomized, Single-blinded Evaluation
Brief Title: Study of the Functional Effects of Nusinersen in 5q-spinal Muscular Amyotrophy Adults (SMA Type 2 or 3 Forms)
Acronym: NUSI-AD-5qSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PO20136
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Spinal Muscular Atrophy
Keywords: oligonucleotides; survival of motor 2 protein; muscular atrophy; quality of life; genetic therapy; single-case studies as topic; humans; adult
MeSH Terms: conditions — Muscular Atrophy, Spinal; Muscular Atrophy | interventions — nusinersen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5q-SMA type 2 and type 3 adults (Experimental): 5q-SMA type 2 and type 3 adults
  Interventions: Other: Monthly assessments of functional motor abilities by a trained therapist; Drug: Nusinersen

INTERVENTIONS:
Other: Monthly assessments of functional motor abilities by a trained therapist — Monthly assessments of functional motor abilities in adult 5q-SMA type 2 and type 3 patients by a trained therapist
Drug: Nusinersen — nusinersen

SUMMARY:
Spinal Muscular Atrophy (SMA) is an autosomal recessive disease caused by a mutation of exon 7, in 95% of cases, encoding the gene for the motor neuron survival protein called SMN1 (Survival Motor Neuron) located on chromosome 5q. Patients with an SMA-5q mutation suffer from progressive muscle deficiency and subsequent atrophy induced by degeneration of motor neurons in the spinal cord. Gene therapy is now available for the management of spinal muscular atrophy and nusinersen is the first approved treatment. Nusinersen has been granted marketing authorization in France since May 30, 2017. Nusinersen has a high level of medical service rendered (MSR) for types I, II, and III, but the improvement in medical service rendered (IMSR) is assessed as moderate for types I and II. For Type III, IMSR is not known.

DETAILED DESCRIPTION:
The aim of the study will be to evaluate the impact on functional motor abilities of intrathecally-injected nusinersen in adult 5q-SMA type 2 and type 3 persons.

If the efficacy of nusinersen protocol will demonstrate the positive impact for patient's, the results of this study would promote an improvement in the medical service rendered in this population in terms of disease stabilization, maintenance of functional capacities and social participation.

ELIGIBILITY:
inclusion criteria :

* Adults (over 18 years of age)
* 5q-SMA type 2 or 3
* with indication for nusinersen treatment by the physician of the center of reference and competence for neuromuscular diseases
* accepting treatment by nusinersen
* Agreeing to participate in the study (signature of the informed consent form).
* living within a radius of 40 km of the investigation center (for logistical reasons related to the conduct of assessments in the patient's home).
* affiliated to a social security system.

exclusion criteria :

* minors (less than 18 years of age)
* with a contra-indication to the nusinersen: pregnancy, breast feeding, hypersensitivity to the nusinersen
* with a contraindication to lumbar puncture: hemostasis disorder, intracerebral mass
* benefiting from another gene therapy drug to treat spinal muscular atrophy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
functional motor ability | 19 months
  functional motor abilities will be evaluate using the Motor Function Measure global score.
  The Motor Function Measure is composed of 32 items, sides from 0 to 3. A high score indicates a better motor function, which can reach a maximum of 96 points.
  The average duration of the test is about 40 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France